CLINICAL TRIAL: NCT01384916
Title: Holistic Approaches to Depression
Acronym: HAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NR012005; 1R01NR012005-01A1 (NIH)
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Depression
Keywords: depression; yoga; health education; antidepressant
MeSH Terms: conditions — Depression; Health Education | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yoga (Experimental)
  Interventions: Behavioral: Yoga
- Health education (Active Comparator)
  Interventions: Behavioral: Healthy Living Workshop

INTERVENTIONS:
Behavioral: Yoga — 2x weekly
  Arms: Yoga
Behavioral: Healthy Living Workshop — 2x weekly
  Arms: Health education

SUMMARY:
The purpose of the study is to investigate whether yoga or a health education group alleviate depressive symptoms for an individual with a partial response to antidepressant medication.

ELIGIBILITY:
Inclusion Criteria:

1. Meets criteria for major depressive disorder (MDD) within the past two years; no history of bipolar disorder, schizophrenia, or psychotic symptoms in one's lifetime.
2. No current hazardous drug/ alcohol use.
3. Depression symptom severity. Participants must have a Quick Inventory of Depressive Symptoms (QIDS) score greater than or equal to 8 and less than or equal to 17.
4. Benefit from current treatment. Participants must report at least some benefit from their current antidepressant.
5. No significant suicidality, defined by a QIDS item #12 score < 2 or PI judgement.
6. Currently taking an antidepressant for depression, at a minimally therapeutic dose. Participant has been taking an antidepressant for at least 8 weeks.
7. Antidepressant dose has not changed in the 4 weeks prior to study entry; Not planning to change antidepressant dosage in next 10 weeks.
8. (If in psychotherapy). Therapist and therapy frequency has not changed in the past 6 weeks AND not planning to change it in the next 3 months.
9. Medically cleared for moderate exercise, documented by a note from their primary care provider.
10. Not pregnant or planning on becoming pregnant in the next year.
11. Naïve to study interventions. Participants cannot have had > 4 single sessions (or > 8 total hours class time) of yoga, other classes in "mindful exercise," (e.g., qigong, tai chi), mindfulness based stress reduction, or health education in the past year or >8 single classes of yoga within the past 2 years of the same. Participants can not have practiced yoga at least once per week for 8 weeks in a row in the past 5 years.
12. Does not practice meditation at home weekly or more often.
13. Understands English sufficiently well to complete study assessment.
14. Biomarker exclusions. Participants who are taking oral steroids, insulin or oral hypoglycemic agents, or oral antibiotics, or who refuse blood draws, will not participate in the biomarker component of the study; however, they may participate in the rest of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2011-06; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptoms (QIDS) | End of acute phase (10 weeks)
  Depression

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Uebelacker, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Nugent NR, Brick L, Armey MF, Tyrka AR, Ridout KK, Uebelacker LA. Benefits of Yoga on IL-6: Findings from a Randomized Controlled Trial of Yoga for Depression. Behav Med. 2021 Jan-Mar;47(1):21-30. doi: 10.1080/08964289.2019.1604489. Epub 2019 May 29. PMID 31141465